CLINICAL TRIAL: NCT00305825
Title: A Phase II Study of Letrozole in Combination With Bevacizumab in Patients With Estrogen Receptor- and/or Progesterone Receptor-Positive Unresectable Locally Advanced and/or Metastatic (Stage IV) Breast Cancer
Brief Title: Bevacizumab and Letrozole in Treating Postmenopausal Women With Locally Advanced or Metastatic Breast Cancer That Cannot Be Removed By Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000465198; UCSF-037518; UCSF-H6961-24611-02; NCT00187694 (obsolete NCT alias)
Record Dates: First submitted 2006-03-21; First posted 2006-03-22 (Estimated); Last update posted 2017-08-31 (Actual); Status verified 2017-08

CONDITIONS: Breast Cancer
Keywords: recurrent breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; stage IV breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Bevacizumab; Letrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Study intervention (Experimental): Patients receive bevacizumab IV over 30-90 minutes on day 1 and oral letrozole once daily on days 1-21. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: bevacizumab; Drug: letrozole

INTERVENTIONS:
Biological: bevacizumab
Drug: letrozole

SUMMARY:
RATIONALE: Monoclonal antibodies, such as bevacizumab, can block tumor growth in different ways. Some find tumor cells and kill them or carry tumor-killing substances to them. Others interfere with the ability of tumor cells to grow and spread. Bevacizumab may also stop the growth of tumor cells by blocking blood flow to the tumor. Estrogen can cause the growth of breast cancer cells. Hormone therapy using letrozole may fight breast cancer by lowering the amount of estrogen the body makes. Giving bevacizumab together with letrozole may be an effective treatment for locally advanced or metastatic breast cancer.

PURPOSE: This phase II trial is studying how well giving bevacizumab together with letrozole works in treating postmenopausal women with locally advanced or metastatic breast cancer that cannot be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the safety and feasibility of bevacizumab in combination with letrozole in postmenopausal women with estrogen receptor- and/or progesterone receptor-positive, unresectable, locally advanced or metastatic breast cancer.

Secondary

* Determine the response rate (partial response [PR] and complete response [CR]) in patients treated with this regimen.
* Determine the clinical benefit rate (PR, CR, and stabilization of disease for ≥ 24 weeks) in patients treated with this regimen.
* Determine the time to progression in patients treated with this regimen.
* Determine the duration of response in patients treated with this regimen.
* Determine the proportion of patients treated with this regimen who have stable disease for ≥ 24 weeks.
* Determine the molecular profile of the patient's breast tumor and explore the relationship between these molecular characteristics and response or resistance to treatment.
* Obtain serial measurements (pre- and post-treatment) of circulating endothelial cells and epithelial cells and explore the relationship between these cells and serum markers of angiogenesis and response to treatment.

OUTLINE: This is a multicenter study.

Patients receive bevacizumab IV over 30-90 minutes on day 1 and oral letrozole once daily on days 1-21. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

PROJECTED ACCRUAL: A total of 42 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed carcinoma of the breast

  * Locally advanced or metastatic (stage IV) disease
  * Unresectable disease
* Measurable or nonmeasurable disease
* May have had stable or progressive disease after ≤ 2 prior conventional chemotherapy regimens for treatment of locally advanced or metastatic breast cancer

  * Prior chemotherapy in the adjuvant or metastatic setting is not required
  * Any number of prior neoadjuvant or adjuvant chemotherapy regimens allowed
  * Prior treatment with high-dose chemotherapy and autologous stem cell or bone marrow transplantation is considered 1 regimen when administered for metastatic disease (including induction chemotherapy and preparative regimen)
* May have had stable or responding disease on prior nonsteroidal aromatase inhibitors (e.g., letrozole, anastrozole, or aminogluthemide)

  * Any prior aromatase inhibitor-related toxicity ≥ grade 3 must have resolved ≥ 4 weeks before the start of study treatment
* May have had disease progression on other prior hormonal therapy (e.g., selective estrogen receptor modulators [SERMs], receptor downregulators [SERDs], or ovarian suppression) in the adjuvant or metastatic setting
* No history or evidence of primary brain tumor or brain metastases by CT scan or MRI
* Must have estrogen receptor- and/or progesterone receptor-positive tumor

PATIENT CHARACTERISTICS:

* Rendered postmenopausal with ovarian suppression (ovarian suppression with a depot LH-RH agonist allowed) prior to the start of study treatment OR is already postmenopausal, as defined by 1 of the criteria:

  * No spontaneous menses for ≥ 12 months if the patient is ≥ 50 years old
  * Amenorrheic for ≥ 12 months if the patient is < 50 years old, with serum estradiol and follicle-stimulating hormone (FSH) levels within the institutional postmenopausal range
  * Bilateral oophorectomy

    * At least 28 days since surgical oophorectomy
  * Patients who have had prior hysterectomy but intact ovaries must be ≥ 55 years old, or have serum estradiol and FSH levels within the postmenopausal range
  * Ongoing ovarian suppression with a depot LH-RH agonist
* ECOG performance status (PS) 0-2 OR Karnofsky PS 60-100%
* Life expectancy > 3 months
* Female only
* Absolute neutrophil count ≥ 1,000/mm^3
* Platelet count ≥ 75,000/mm^3
* WBC ≥ 2,500/mm^3
* AST and ALT ≤ 2.5 times upper limit of normal
* Bilirubin normal
* Creatinine normal OR creatinine clearance ≥ 60 mL/min
* No proteinuria at baseline

  * Patients who unexpectedly have ≥ +1 proteinuria must undergo a 24-hour urine collection that demonstrates ≤ 500 mg of protein over 24 hours
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No presence of bleeding diathesis or coagulopathy
* No history of allergic reaction to compounds of similar chemical or biologic composition to letrozole or bevacizumab
* No serious, nonhealing wound, ulcer, or bone fracture
* No unstable angina pectoris
* No serious cardiac arrhythmia requiring medication
* No uncontrolled hypertension
* No myocardial infarction
* No New York Heart Association class II-IV congestive heart failure
* No peripheral vascular disease ≥ grade II within the past year
* No other clinically significant cardiovascular disease
* No history or evidence of other CNS disease by CT scan or MRI, including seizures not controlled with standard medical therapy or stroke
* No gastrointestinal tract disease resulting in an inability to take oral medication
* No requirement for IV alimentation
* No significant traumatic injury within the past 28 days
* No psychiatric illness or social situation that would preclude study compliance
* No other uncontrolled intercurrent illness

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior steroidal aromatase inhibitors (e.g., exemestane) unless administered in the adjuvant setting (not for metastatic disease) and ≥ 12 months have elapsed since last treatment
* Any number of prior immunotherapies (e.g., trastuzumab [Herceptin^®] or vaccines) in the adjuvant or metastatic setting allowed
* More than 3 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin C)
* More than 3 weeks since prior radiotherapy
* More than 3 weeks since prior immunotherapy
* More than 3 weeks since prior investigational therapy
* More than 2 weeks since prior hormonal therapy except letrozole therapy or a luteinizing hormone-releasing hormone (LH-RH) agonist for ovarian suppression
* No prior surgical procedures affecting absorption
* More than 28 days since prior major surgery or open biopsy
* At least 24 hours since prior placement of indwelling catheters
* At least 10 days since prior and no concurrent full-dose oral or parenteral anticoagulants or thrombolytic agents except as required to maintain patency of preexisting, permanent indwelling IV catheters

  * Patients receiving warfarin should have INR < 1.5
* No prior bevacizumab
* No other prior KDR inhibitors (e.g., vascular endothelial growth factor [VEGF] Trap, SU5416, SU6668, ZD6474, vatalanib, AEE788, or IMC-1CII)
* No other concurrent investigational agent
* No concurrent chronic daily treatment with aspirin (> 325 mg/day) or nonsteroidal anti-inflammatory medications known to inhibit platelet function (e.g., cyclooxygenase-1 inhibitors)
* Concurrent bisphosphonates (e.g., zoledronate or pamidronate) or growth factors allowed
* No other concurrent anticancer agents or therapies

Ages: 18 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2004-08; Primary Completion 2006-05-30 (Actual); Study Completion 2016-05-24 (Actual)

PRIMARY OUTCOMES:
Safety
Feasibility

SECONDARY OUTCOMES:
Response rate (complete response and partial response)
Clinical benefit rate (complete response, partial response, and stable disease for at least 24 weeks)
Time to progression
Duration of response

CONTACTS AND LOCATIONS:
Overall Officials: Hope S. Rugo, MD, Principal Investigator — University of California, San Francisco
Locations (2):
- United States (2):
  - UCSF Comprehensive Cancer Center, San Francisco, California
  - Memorial Sloan-Kettering Cancer Center, New York, New York

REFERENCES:
- [Result] Traina TA, Rugo HS, Caravelli JF, Patil S, Yeh B, Melisko ME, Park JW, Geneus S, Paulson M, Grothusen J, Seidman AD, Fornier M, Lake D, Dang C, Robson M, Theodoulou M, Flombaum CD, Norton L, Hudis CA, Dickler MN. Feasibility trial of letrozole in combination with bevacizumab in patients with metastatic breast cancer. J Clin Oncol. 2010 Feb 1;28(4):628-33. doi: 10.1200/JCO.2009.21.8784. Epub 2009 Oct 19. PMID 19841327